CLINICAL TRIAL: NCT05593991
Title: Immediate Repercussions on the Spine Posture From Passive Elevation of the Heels in Healthy Subjects: a Cross-sectional Study
Brief Title: Immediate Repercussions of High Heels on Spine Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manusapiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H&S01
Record Dates: First submitted 2022-10-13; First posted 2022-10-26 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adults (Experimental): Subjects with elevated heels
  Interventions: Other: Elevated heels

INTERVENTIONS:
Other: Elevated heels — Each subject will undergo the following evaluations:
  1. neutral barefoot position;
  2. neutral barefoot position (re-test);
  3. 3 cm rise of both heels, made with plastic spacer;
  4. 7 cm rise of both heels, made with plastic spacer.

SUMMARY:
The goal of this cross-sectional study is to evaluate the immediate effect of heels elevation on the spine posture in a group of 100 healthy subjects (50 males, 50 females). The main question it aims to answer is weather high heels immediately affects spinal posture and pelvic position in the sagittal plane.

Participants will undergo an elevation of 3cm and then 7cm of both heels, while their spine posture will be examined by means of a rasterstereography device.

DETAILED DESCRIPTION:
The data collected by the rasterstereography device will be:

1. pelvic tilt angle (PI), the angle determined by the vertical and the tangent to lumbosacral junction (ILS);
2. ITL-ILS lordotic angle, measured between the tangents of the thoracolumbar junction (ITL) and the lumbosacral junction (ILS);
3. ICT-ITL kyphotic angle, measured between the tangents of the cervicothoracic junction (ICT) and the thoracolumbar junction (ITL); see fig. 1;
4. lumbar arrow (FL) horizontal distance in millimeters from the vertical line that passes through the kyphotic apex in the lumbar spine;
5. cervical arrow (FC) (horizontal distance in millimeters from the virtual vertical plumb line that passes through the kyphotic apex in the cervical spine);
6. antero-posterior flexion of the trunk (Trunk Inclination-TI) measured as the angle between the vertical line and the line passing through the prominent cervical vertebra (VP) to the line connecting the two dimples (DM); see fig. 2.

Participants will provide information on age, height and weight. A questionnaire will be administered to standardize the types of high-heeled shoes used and to verify their frequency of use.

Evaluation Protocol

1. sample 1: barefoot neutral position;
2. sample 2: barefoot neutral position;
3. sample 3: 3 cm rise under both heels;
4. sample 4: 7 cm rise under both heels.

The positioning with respect to the measurement system will be carried out according to the indications provided by the supplier.

To standardize the position subjects will be prepared for analysis as follows:

1. standing, back to the detection system, in a relaxed posture with the knees fully extended with bare feet on the floor (neutral position);
2. bare trunk with pants and briefs lowered to half of the glutei
3. in the case of long hair, it will be required to tie it with suitable means (cap, hair clips, hair bands, etc.) so that the neck is visible up to the hairline;
4. rings, watches and necklaces will be removed to avoid any interference with light lines (necklaces in particular increase this probability).

In the third survey, the heel will be raised by inserting a plastic bar symmetrically under both heels, as proposed in previous studies in which wood was used, by 3 cm; for the fourth evaluation it will be 7 cm.

After the first evaluation in the neutral position, before the evaluation with the heel lift, a second evaluation will be performed under the same conditions to evaluate the reproducibility of the data. The time between the two assessments will be less than 1 minute and the subject will not change position.

ELIGIBILITY:
Inclusion Criteria:

All healthy subjects.

Exclusion Criteria:

* structural or neurological abnormalities that would prevent standing for 5 seconds with their heels on a 7 cm high plinth;
* regular users of shoes with 7 cm high heels (or more), with a frequency of more than twice a week and / or more than 3 hours / week;
* low back pain in the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
pelvic tilt angle | 5 seconds for each measured condition (barefoot, 3 cm heels elevation, 7 cm heels elevation)
  the angle between the vertical and the tangent to the lumbosacral junction
lordotic angle | 5 seconds for each measured condition (barefoot, 3 cm heels elevation, 7 cm heels elevation)
  measured between the tangents of the thoracolumbar junction and the lumbosacral junction;
kyphotic angle | 5 seconds for each measured condition (barefoot, 3 cm heels elevation, 7 cm heels elevation)
  measured between the tangents of the cervicothoracic junction and the thoracolumbar junction;
lumbar arrow | 5 seconds for each measured condition (barefoot, 3 cm heels elevation, 7 cm heels elevation)
  horizontal distance in millimeters of the lumbar spine from the virtual vertical line that passes through the kyphotic apex;
cervical arrow | 5 seconds for each measured condition (barefoot, 3 cm heels elevation, 7 cm heels elevation)
  horizontal distance in millimeters of the cervical spine from the virtual vertical line that passes through the kyphotic apex;
anteroposterior trunk flexion | 5 seconds for each measured condition (barefoot, 3 cm heels elevation, 7 cm heels elevation)
  measured as the angle between the vertical and the line that passes through the prominent cervical vertebra and the line connecting the two dimples.

CONTACTS AND LOCATIONS:
Overall Officials: Saverio Colonna, MD, Principal Investigator — Spine Center
Locations (1):
- Spine Center, Bologna, Italy

REFERENCES:
- [Background] Bird AR, Bendrups AP, Payne CB. The effect of foot wedging on electromyographic activity in the erector spinae and gluteus medius muscles during walking. Gait Posture. 2003 Oct;18(2):81-91. doi: 10.1016/s0966-6362(02)00199-6. PMID 14654211
- [Background] Snow RE, Williams KR. High heeled shoes: their effect on center of mass position, posture, three-dimensional kinematics, rearfoot motion, and ground reaction forces. Arch Phys Med Rehabil. 1994 May;75(5):568-76. PMID 8185452
- [Background] Cowley EE, Chevalier TL, Chockalingam N. The effect of heel height on gait and posture: a review of the literature. J Am Podiatr Med Assoc. 2009 Nov-Dec;99(6):512-8. doi: 10.7547/0990512. PMID 19917737
- [Background] de Oliveira Pezzan PA, Joao SM, Ribeiro AP, Manfio EF. Postural assessment of lumbar lordosis and pelvic alignment angles in adolescent users and nonusers of high-heeled shoes. J Manipulative Physiol Ther. 2011 Nov;34(9):614-21. doi: 10.1016/j.jmpt.2011.09.006. PMID 22078999
- [Background] Dai M, Li X, Zhou X, Hu Y, Luo Q, Zhou S. High-heeled-related alterations in the static sagittal profile of the spino-pelvic structure in young women. Eur Spine J. 2015 Jun;24(6):1274-81. doi: 10.1007/s00586-015-3857-6. Epub 2015 Mar 10. PMID 25753007
- [Background] de Lateur BJ, Giaconi RM, Questad K, Ko M, Lehmann JF. Footwear and posture. Compensatory strategies for heel height. Am J Phys Med Rehabil. 1991 Oct;70(5):246-54. PMID 1910649
- [Background] Franklin ME, Chenier TC, Brauninger L, Cook H, Harris S. Effect of positive heel inclination on posture. J Orthop Sports Phys Ther. 1995 Feb;21(2):94-9. doi: 10.2519/jospt.1995.21.2.94. PMID 7711763
- [Background] Bendix T, Sorensen SS, Klausen K. Lumbar curve, trunk muscles, and line of gravity with different heel heights. Spine (Phila Pa 1976). 1984 Mar;9(2):223-7. doi: 10.1097/00007632-198403000-00016. PMID 6729584
- [Background] Chodick G, Ronckers CM, Shalev V, Ron E. Excess lifetime cancer mortality risk attributable to radiation exposure from computed tomography examinations in children. Isr Med Assoc J. 2007 Aug;9(8):584-7. PMID 17877063
- [Background] Drerup B, Ellger B, Meyer zu Bentrup FM, Hierholzer E. [Functional rasterstereographic images. A new method for biomechanical analysis of skeletal geometry]. Orthopade. 2001 Apr;30(4):242-50. doi: 10.1007/s001320050603. German. PMID 11357446
- [Background] Opila KA, Wagner SS, Schiowitz S, Chen J. Postural alignment in barefoot and high-heeled stance. Spine (Phila Pa 1976). 1988 May;13(5):542-7. doi: 10.1097/00007632-198805000-00018. PMID 3187700

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT05593991/Prot_SAP_000.pdf